CLINICAL TRIAL: NCT07000123
Title: A Phase III, Randomised, Double-Blind, Placebo-Controlled, Parallel-Group Study to Assess the Effect of AZD0780 on Low-Density Lipoprotein Cholesterol in Patients With Elevated Low Density Lipoprotein Cholesterol and Clinical Atherosclerotic Cardiovascular Disease or at Risk for a First Atherosclerotic Cardiovascular Disease Event
Brief Title: A Phase III Study to Assess the Effect of AZD0780 on LDL-C in Patients With Clinical ASCVD or at Risk for a First ASCVD Event
Acronym: AZURE-LDL
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D7960C00012; 2025-520521-21 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2025-05-23; First posted 2025-06-02 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Cardiovascular Disease
Keywords: Low-Density Lipoprotein Cholesterol; Atherosclerotic Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis

STUDY DESIGN:
Intervention Model Description: International, multi-centre, randomised, double-blind, placebo-controlled, parallel-group
Who Masked: Participant, Care Provider, Investigator
Masking Description: Placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AZD0780 (Experimental): Participants will receive daily oral dose of AZD0780
  Interventions: Drug: AZD0780
- Placebo (Placebo Comparator): Participants will receive daily oral dose of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD0780 — Participants will receive daily oral dose of AZD0780
  Arms: AZD0780
Drug: Placebo — Participants will receive daily oral dose of placebo
  Arms: Placebo

SUMMARY:
This is a study to evaluate the efficacy and safety of AZD0780 in adults with clinical ASCVD or who are at risk for a first ASCVD event and who have elevated LDL-C. AZD0780 is a small molecule that reduces the amount of LDL-C in the blood. Placebo will be used for comparison, and neither the participants nor the Investigators will know who is receiving the AZD0780 medication and who is receiving the placebo until the end of study.

The total length of the study for an individual participant will be up to approximately 56 weeks, including a screening period of up to 14 days, treatment with AZD0780 or placebo for 52 weeks, and a safety follow-up period of 10 days.

DETAILED DESCRIPTION:
This is a randomised, double-blind, placebo-controlled, parallel-group Phase III study to evaluate the effect on the reduction of LDL-C and the safety and tolerability of AZD0780 versus placebo, administered as xx mg once daily orally, on top of a high intensity lipid-lowering regimen. The target population is adults ≥ 18 years of age with LDL-C ≥ 55 mg/dL and history of clinical ASCVD or ≥ 70 mg/dL and at risk for a first ASCVD event.

The study will be conducted at approximately 470 centres in approximately 21 countries.

The screening period is up to 14 days (and may be conditionally extended), starts at the date of signed informed consent, and ends on the day before the randomisation visit. Participants will be randomised in a 1:1 ratio to either AZD0780 or placebo for a treatment period of 52 weeks and a 10-day safety follow-up. Those randomised to the AZD0780 group will receive AZD0780 xx mg orally once daily during the treatment period, while those in the placebo group will receive matching placebo. The study will include approximately 2800 randomised participants. An independent data monitoring committee will, on a regular basis, review accumulating data from the study, evaluate adverse effects of the IMP, and make recommendations regarding whether to halt or modify the study.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age at the time of signing the ICF
* History of clinical ASCVD or at risk for a first ASCVD event:

  1. Clinical ASCVD is defined as MI, stable or unstable angina, coronary or other arterial revascularisation, ischaemic stroke, or peripheral artery disease.
  2. A participant is considered at risk for a first ASCVD event if the participant has one or more of the following conditions: atherosclerotic vascular disease (≥ 50% stenosis in ≥ 2 coronary artery territories or in ≥ 2 vascular beds [coronary, carotid, lower extremity], diagnosed by any imaging modality), diabetes mellitus, hypertension, cigarette smoking, chronic kidney disease (moderate to severe stage), or obesity. Investigators can also use the ACC/AHA or ESC or other relevant national clinical guidelines for risk assessment to identify participants with at least moderate risk for ASCVD.
* Fasting serum LDL-C by central laboratory at screening as follows: LDL-C ≥ 55 mg/dL (≥ 1.4 mmol/L) in participants with clinical ASCVD or ≥ 70 mg/dL (≥ 1.8 mmol/L) in participants without clinical ASCVD but at risk for a first ASCVD event
* Participants should receive a background lipid lowering regimen anticipated to achieve at least a ~50% reduction in LDL-C. Except in cases of intolerance, the regimen should include a high intensity statin therapy or lower intensity statin therapy in combination with an oral agent with proven outcome benefit (eg, ezetimibe and/or bempedoic acid).

Thus, the background lipid-lowering therapy must consist of one of the following:

- A high intensity LDL lowering regimen

(i) A high intensity statin regimen, as defined by country specific guidelines OR: (ii) A lower intensity statin regimen in combination with ezetimibe and/or bempedoic acid :

OR:

- A maximum tolerated statin regimen - Oral combination therapy with ezetimibe and/or bempedoic acid is strongly recommended.

Participants must achieve a stable background lipid lowering therapy > 28 days before screening.

Exclusion criteria:

* Homozygous familial hypercholesterolaemia, known diagnosis of HeFH, LDL apheresis or plasma apheresis within 12 months prior to screening, or any other underlying known disease or condition that may interfere with interpretation of the clinical study results as judged by the Investigator.
* Any of the following laboratory values at screening:

  * Calculated eGFR < 15 mL/min/1.73 m2
  * AST or ALT > 3 × ULN
  * TBL > 2 × ULN (except for patients with Gilberts syndrome, where TBL 3 × ULN is acceptable provided direct bilirubin < 1.5 × ULN)
  * Fasting triglycerides ≥ 400 mg/dL (≥ 4.52 mmol/L)
  * Creatine kinase > 5 × ULN
  * Urine albumin-to-creatinine ratio ≥ 500 mg/g
* Uncontrolled type 2 diabetes mellitus defined as HbA1C ≥ 9.5% at screening
* Inadequately treated hypothyroidism defined as TSH > 1.5 ULN at screening or participants whose thyroid replacement therapy was initiated or modified within the last 3 months prior to screening
* Use of mipomersen or lomitapide (cholesterol-lowering medications) within 12 months prior to screening or planned use during the study.
* Use of gemfibrozil within 1 week prior to screening or planned use during the study.
* Use of PCSK-9 inhibitors: evolocumab/alirocumab within 12 weeks of the screening visit or planned use during the study or inclisiran within 18 months of the screening visit or planned use during the study. Any other approved PCSK-9 inhibitor use within 5 half-lives prior to the screening visit or planned use during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3046 (Actual)
Dates: Start 2025-05-28 (Actual); Primary Completion 2027-01-11 (Estimated); Study Completion 2027-01-11 (Estimated)

PRIMARY OUTCOMES:
Relative change in LDL-C from baseline to 12 weeks | Baseline - 12 weeks
  To compare the effect of treatment with AZD0780 versus placebo on LDL-C at 12 weeks

SECONDARY OUTCOMES:
Relative change in LDL-C from baseline to 12 weeks | Baseline - 12 weeks
  To compare the effect of treatment with AZD0780 versus placebo on LDL-C at 12 weeks in patients on background statin therapy
Indicator for LDL-C < 70 mg/dL (< 1.8 mmol/L) at 12 weeks | Baseline - 12 weeks
  To compare the effect of treatment with AZD0780 versus placebo on the probability of LDL-C < 70 mg/dL at 12 weeks in patients with baseline LDL-C ≥ 70 mg/dL
Indicator for LDL-C < 55 mg/dL (< 1.4 mmol/L) at 12 weeks | Baseline - 12 weeks
  To compare the effect of treatment with AZD0780 versus placebo on the probability of LDL-C < 55 mg/dL at 12 weeks
Relative change in LDL-C from baseline to 28 weeks | Baseline - 28 weeks
  To compare the effect of treatment with AZD0780 versus placebo on LDL-C at 28 weeks
Relative change in LDL-C from baseline to 52 weeks | Baseline - 52 weeks
  To compare the effect of treatment with AZD0780 versus placebo on LDL-C at 52 weeks
Relative change in Apo B from baseline to 12 weeks | Baseline - 12 weeks
  To compare the effect of treatment with AZD0780 versus placebo on apolipoprotein (Apo) B at 12 weeks
Relative change in non-HDL-C from baseline to 12 weeks | Baseline - 12 weeks
  To compare the effect of treatment with AZD0780 versus placebo on non-high-density lipoprotein cholesterol (HDL-C) at 12 weeks
Relative change in total cholesterol from baseline to 12 weeks | Baseline - 12 weeks
  To compare the effect of treatment with AZD0780 versus placebo on total cholesterol at 12 weeks
Relative change in Lp(a) from baseline to 12 weeks | Baseline - 12 weeks
  To compare the effect of treatment with AZD0780 versus placebo on lipoprotein(a) (Lp[a]) at 12 weeks

CONTACTS AND LOCATIONS:
Locations (321):
- United States (95):
  - Research Site, Huntsville, Alabama
  - Research Site, Irondale, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Gilbert, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Sun City West, Arizona
  - Research Site, Garden Grove, California
  - Research Site, Gardena, California
  - Research Site, Lancaster, California
  - Research Site, Lincoln, California
  - Research Site, San Diego, California
  - Research Site, Torrance, California
  - Research Site, West Hills, California
  - Research Site, Hamden, Connecticut
  - Research Site, Boca Raton, Florida
  - Research Site, Hallandale, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Inverness, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, New Port Richey, Florida
  - Research Site, Orlando, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Seminole, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Decatur, Georgia
  - Research Site, Peachtree Corners, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Winfield, Illinois
  - Research Site, Evansville, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, Ames, Iowa
  - Research Site, El Dorado, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Owensboro, Kentucky
  - Research Site, Hammond, Louisiana
  - Research Site, Kenner, Louisiana
  - Research Site, Lafayette, Louisiana
  - Research Site, Lake Charles, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Zachary, Louisiana
  - Research Site, Annapolis, Maryland
  - Research Site, Baltimore, Maryland
  - Research Site, Beltsville, Maryland
  - Research Site, Potomac, Maryland
  - Research Site, Chesterfield, Missouri
  - Research Site, Jefferson City, Missouri
  - Research Site, Kansas City, Missouri
  - Research Site, Missoula, Montana
  - Research Site, Buffalo, New York
  - Research Site, Rochester, New York
  - Research Site, The Bronx, New York
  - Research Site, Durham, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Hickory, North Carolina
  - Research Site, Morganton, North Carolina
  - Research Site, New Bern, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Rocky Mount, North Carolina
  - Research Site, Salisbury, North Carolina
  - Research Site, Statesville, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Blue Ash, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Lima, Ohio
  - Research Site, Camp Hill, Pennsylvania
  - Research Site, Horsham, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, West Chester, Pennsylvania
  - Research Site, Anderson, South Carolina
  - Research Site, Fort Mill, South Carolina
  - Research Site, Mauldin, South Carolina
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, North Charleston, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Bristol, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Beaumont, Texas
  - Research Site, El Paso, Texas
  - Research Site, Houston, Texas
  - Research Site, Humble, Texas
  - Research Site, Irving, Texas
  - Research Site, Katy, Texas
  - Research Site, Mesquite, Texas
  - Research Site, Paris, Texas
  - Research Site, San Antonio, Texas
  - Research Site, San Marcos, Texas
  - Research Site, Sugar Land, Texas
  - Research Site, Charlottesville, Virginia
  - Research Site, Hampton, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Suffolk, Virginia
  - Research Site, Redmond, Washington
- Argentina (10):
  - Research Site, CABA
  - Research Site, Ciudad Autonoma de Bs As
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Córdoba
  - Research Site, Godoy Cruz
  - Research Site, Mar del Plata
  - Research Site, Rosario
  - Research Site, San Nicolás
  - Research Site, San Vicente
  - Research Site, Zárate
- Australia (8):
  - Research Site, Coffs Harbour
  - Research Site, Ipswich
  - Research Site, Joondalup
  - Research Site, Leabrook
  - Research Site, Liverpool
  - Research Site, Maroubra
  - Research Site, Melbourne
  - Research Site, Woolloongabba
- Brazil (7):
  - Research Site, Brasília
  - Research Site, Campina Grande do Sul
  - Research Site, Campinas
  - Research Site, Goiânia
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, São Paulo
- Bulgaria (6):
  - Research Site, Dupnitsa
  - Research Site, Haskovo
  - Research Site, Plovdiv
  - Research Site, Sliven
  - Research Site, Sofia
  - Research Site, Varna
- Canada (17):
  - Research Site, Surrey, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research Site, Cambridge, Ontario
  - Research Site, Courtice, Ontario
  - Research Site, Guelph, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, North York, Ontario
  - Research Site, Sarnia, Ontario
  - Research Site, Stoney Creek, Ontario
  - Research Site, Stouffville, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Chicoutimi, Quebec
  - Research Site, Joliette, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Sherbrooke, Quebec
- Chile (4):
  - Research Site, Independencia
  - Research Site, Santiago
  - Research Site, Valdivia
  - Research Site, Victoria
- Czechia (13):
  - Research Site, Benešov
  - Research Site, Brandýs nad Labem
  - Research Site, Chlumec nad Cidlinou
  - Research Site, České Budějovice
  - Research Site, Hodonín
  - Research Site, Jílové u Prahy
  - Research Site, Klatovy
  - Research Site, Prague
  - Research Site, Praha Uhříněves
  - Research Site, Příbram
  - Research Site, Teplice
  - Research Site, Trutnov
  - Research Site, Uherské Hradiště
- Germany (31):
  - Research Site, Amberg
  - Research Site, Bad Homburg
  - Research Site, Berlin
  - Research Site, Dresden
  - Research Site, Essen
  - Research Site, Falkensee
  - Research Site, Frankfurt
  - Research Site, Freiburg im Breisgau
  - Research Site, Greifswald
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Hohenmölsen
  - Research Site, Kaiserslautern
  - Research Site, Karlsruhe
  - Research Site, Kiel
  - Research Site, Leipzig
  - Research Site, Magdeburg
  - Research Site, Mannheim
  - Research Site, Markkleeberg
  - Research Site, Munich
  - Research Site, München
  - Research Site, Münster
  - Research Site, Nuremberg
  - Research Site, Offenbach
  - Research Site, Potsdam
  - Research Site, Schwerin
  - Research Site, Stuhr
  - Research Site, Stuttgart
  - Research Site, Wermsdorf
  - Research Site, Witten
- Hungary (14):
  - Research Site, Balatonfüred
  - Research Site, Békéscsaba
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Dunaújváros
  - Research Site, Kalocsa
  - Research Site, Kaposvár
  - Research Site, Nyíregyháza
  - Research Site, Nyíregyháza-Sóstóhegy
  - Research Site, Orosháza
  - Research Site, Pécs
  - Research Site, Szeged
  - Research Site, Székesfehérvár
  - Research Site, Zalaegerszeg
- India (5):
  - Research Site, Belagavi
  - Research Site, Dehradun
  - Research Site, Kanpur
  - Research Site, Kochi
  - Research Site, New Delhi
- Japan (22):
  - Research Site, Ami-machi
  - Research Site, Asahi-shi
  - Research Site, Chūōku
  - Research Site, Hamamatsu
  - Research Site, Ichikawa-shi
  - Research Site, Kanazawa
  - Research Site, Kasuya-gun
  - Research Site, Kishiwada-shi
  - Research Site, Kitakyushu
  - Research Site, Komatsu-shi
  - Research Site, Kure-shi
  - Research Site, Minatoku
  - Research Site, Nagoya
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Suwa-shi
  - Research Site, Tamanashi
  - Research Site, Tsukuba
  - Research Site, Urasoe-Shi
  - Research Site, Ushiku-shi
  - Research Site, Utsunomiya
  - Research Site, Yokohama
- Malaysia (7):
  - Research Site, Bandar Aman Jaya
  - Research Site, Ipoh
  - Research Site, Kuching
  - Research Site, Sarawak Miri
  - Research Site, Seri Manjung
  - Research Site, Sibu
  - Research Site, Sungai Buloh
- Poland (15):
  - Research Site, Bialystok
  - Research Site, Gdansk
  - Research Site, Gdynia
  - Research Site, Katowice
  - Research Site, Kędzierzyn-Koźle
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Poznan
  - Research Site, Płock
  - Research Site, Rzeszów
  - Research Site, Szczecin
  - Research Site, Warsaw
  - Research Site, Wroclaw
  - Research Site, Zabrze
- Slovakia (10):
  - Research Site, Bratislava
  - Research Site, Košice
  - Research Site, Levice
  - Research Site, Lučenec
  - Research Site, Malacky
  - Research Site, Námestovo
  - Research Site, Prešov
  - Research Site, Rožňava
  - Research Site, Svidník
  - Research Site, Vinica
- South Korea (15):
  - Research Site, Anyang-si
  - Research Site, Bucheon-si
  - Research Site, Busan
  - Research Site, Changwon-si
  - Research Site, Cheonan-si
  - Research Site, Daegu
  - Research Site, Daejeon
  - Research Site, Gangwon-do
  - Research Site, Goyang-si
  - Research Site, Gwangju
  - Research Site, Jeju City
  - Research Site, Jeonju
  - Research Site, Jinju
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (6):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, Madrid
  - Research Site, Santiago(A Coruña)
  - Research Site, Seville
- Taiwan (4):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
- Turkey (Türkiye) (8):
  - Research Site, Adana
  - Research Site, Afyonkarahisar
  - Research Site, Ankara
  - Research Site, Eskişehir
  - Research Site, Izmir
  - Research Site, Kocaeli
  - Research Site, Odunpazari
  - Research Site, Yenimahalle
- Ukraine (5):
  - Research Site, Chernivtsi
  - Research Site, Ivano-Frankivsk
  - Research Site, Kyiv
  - Research Site, Lutsk
  - Research Site, Vinnytsia
- United Kingdom (15):
  - Research Site, Chesterfield
  - Research Site, Chippenham
  - Research Site, Corby
  - Research Site, Coventry
  - Research Site, Harrow
  - Research Site, Hull
  - Research Site, London
  - Research Site, Northwood
  - Research Site, Orpington
  - Research Site, Poole
  - Research Site, Rotherham
  - Research Site, Shipley
  - Research Site, Thetford
  - Research Site, Trowbridge
  - Research Site, Weston-super-Mare
- Vietnam (4):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City
  - Research Site, Hochiminh
  - Research Site, Huế

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/